CLINICAL TRIAL: NCT04170699
Title: Effects of Ultrasound Guided Pectoral Blok Type 1 on Subcutaneous Port Catheter Replacement : A Randomized Controlled Study
Brief Title: Effects of PECS 1 Block on Venous Cancer Port Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, OZCAN PISKIN, MD, ASSOCIATED PROFFESOR OZCAN PISKIN M.D., Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-78-08/05
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Catheter; Pain (Indwelling Catheter)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study will be a two-arm parallel assignment. One group will receive PECS 1 block and the other will receive infiltrative anesthesia.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS 1 Block (Experimental): 40 patients who had PECS 1 block for peroperative analgesia in port-a-cath replacement. All patients will receive IV Midazolam (0.05mg/kg) premedication. Standard monitorization of EKG, non- invasive blood pressure and pulseoximeter will be done and recorded in every 5 minutes. After sedation and standard monitorization, 20 minutes before the intervention and in the supine positon the PECS 1 block will be done. 10 % povidone - iodin will be used for sterilization and the USG probe will be covered with sterile sheath. The block will be done as a single injection of local anaesthetic between pectoralis major and pectoralis minor muscles at the level of the 3rd rib to anaesthetise the lateral and medial pectoral nerves. The USG probe will be replaced inferior to the clavicle. Identify the pectoralis muscles with the axillary artery and axillary vein on sonography. The brachial plexus should be visible underneath. After confirmation with 20 mL %0.25 bupivacaine will be administered.
  Interventions: Procedure: Port-a-cath replacement
- Infiltrative Anesthesia (Experimental): 40 patients who had port-cath replacement will receive infiltrative anesthesia.
  Interventions: Procedure: Port-a-cath replacement

INTERVENTIONS:
Procedure: Port-a-cath replacement — Implantation of a subcutaneous venous port-a-cath

SUMMARY:
In this study our aim is to investigate the effects of ultrasound (USG) guided pectoral block (PECS) type 1 in the administration of an implanted port-a-cath .

DETAILED DESCRIPTION:
Cancer is one of the most important reasons of mortality in the world. There are a lot of different types of treatments for cancer and so far chemotherapy is the most common one. However, chemotherapy damages the peripheral veins, so implanted subcutaneous port-a-caths are used as an alternative. Traditionally this implantation is adminstered with infiltrative anesthesia. Recently, USG is used in anesthesia practice world wide. Blanco R et all (1) defined PECS 1 block as an alternative to paravertebral block. PECS 1 block aims to anesthetize the medial and lateral pectoral nerves. In this study our aim is to investigate the effects of USG guided PECS 1 block in the administiration of an implanted port-a-cath .

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18- 75
* ASA (American Society of Anesthesiologists) Score I-IV
* Undergoing elective port-a-cath replacemnet

Exclusion Criteria:

* Patients with neurological deficits
* Patients who have major vascular damage at the same side
* Mentally retarded patients
* Patients with alcohol or drug addiction
* Patients who are allergic to local anesthetics
* Pregnancy
* Paitents with coagulopathy
* Patients with skin infection at the side of the procedure
* Patients with pneumothorax at the side of the procedure
* Patient with a pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Perioperative and postoperative analgesic needs of patients | Change in Visual analog Scale (VAS) scores ( between 1 and 10, a higher score represents greater pain intensity. ) at the 1st, 3rd, 6th, 12th and 24th hours after the procedure.
  Our primary outcome is to measure and identify the analgesic needs of the patients at the perioperative and postoperative period.In order to measure the analgesic needs Visual Analogue Scale will be used and patients' pain scores will be measured.

SECONDARY OUTCOMES:
Hemodynamic parameters at the perioperative and postoperative period | 1st, 3rd, 6th,12th and 24th hours after the procedure.
  Our secondary outcome is to measure the hemodynamic parameters such as systolic and diastolic arterial pressure at the perioperative and postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: OZCAN PISKIN, M.D., Principal Investigator — Bulent Ecevit University
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No